CLINICAL TRIAL: NCT04544930
Title: Therapist-guided Internet Treatment for Hazardous and Harmful Alcohol Use. a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31352
Record Dates: First submitted 2020-07-08; First posted 2020-09-10 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Alcohol Abuse; Internet-Based Intervention
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- therapist-guided (Experimental): Therapist-guided Internet treatment based on cognitive behavior therapy (ICBT).
  Interventions: Behavioral: therapist-guided

INTERVENTIONS:
Behavioral: therapist-guided — Therapist-guided Internet treatment comprises eight text modules on the Internet that include psychoeducation, tasks and exercises. Key elements are setting goals for treatment, identifying and challenging negative automatic thoughts through a number of exercises and behavioral experiments, as well as making a plan for relapse prevention. Therapist guidance is secondary to the self-help modules, and the therapist provides feedback to the patient online in the secured program once a week

SUMMARY:
The aim of the present study is to test the feasibility of therapist-guided Internet treatment for hazardous (risky) and harmful alcohol use among adults 18 years and older. The hypothesis is that the intervention is feasible and that it can help people change risky drinking habits at an early stage before developing into problems that are more serious.The therapist-guided Internet treatment addresses the person's need for confidentiality and contributes to reducing the stigma associated with visiting a substance abuse clinic.

DETAILED DESCRIPTION:
Background:

A significant proportion of people with substance abuse do not seek help for their problems and therefore do not receive the necessary help at an early stage. An important reason for this is the stigma associated with substance abuse. Therapist-guided Internet treatment has been developed and tested in recent years as an approach that increases access to effective treatment for a variety of mental and substance-related problems and disorders. Internet-based interventions increase the patient's choice of type of treatment and give the patient an experience of having control over their own behavior change. Moreover, such treatment is independent of where you live, and you do not need to attend a clinic. In addition, by offering therapist-guided Internet treatment, therapists can treat far more patients compared to regular face-to-face treatment. In this way, the health services, which are already under severe pressure due to many new and competing tasks, are relieved.

Research questions:

1. Is therapist-guided Internet treatment for hazardous and harmful alcohol use feasible for self-referred persons?
2. What factors contribute/do not contribute to the feasibility of treatment?
3. Can the intervention help people change risky drinking habits before it develops into problems that are more serious?
4. How do participants experience the intervention?

Methods:

Participants:

A total of 30 participants will be recruited through announcements in social media, newspapers and through GP's and other health care services. Participants will be recruited from the catchment area of Haukeland University Hospital, Western Norway, and Vestfold Hospital, Eastern Norway.

Design:

The study will be conducted as an open, 6-months follow-up study, to assess whether the design is suitable for a randomized controlled trial in the next round. Both quantitative and qualitative methods will be used to investigate the feasibility of the treatment program.

Data collection:

Assessments will be carried out at start of treatment (T1), through the treatment course (T2) and at the end of treatment (T3) and at follow-up (T4). Qualitative interviews will be conducted at the end of treatment.

Intervention:

The treatment program is developed at Vestfold Hospital, Norway. It is based on Internet- based cognitive behavior therapy (ICBT). The treatment program consists of eight text-based self-help modules on the Internet that participants can access via secure login using Bank identification (ID) (security level 4). The self-help modules include psychoeducation, tasks and exercises. The therapist guidance is secondary to the self-help modules. The therapist provides feedback to the patient online in the secured program once a week.

Statistics:

Sample size:

Since this is a feasibility study primarily intended to test the feasibility of therapist-guided Internet treatment for hazardous and harmful alcohol use, the sample will be limited to 30 participants. Therefore, power analysis is not performed.

Statistical methods:

Both statistical and interpretative methods will be used. Descriptive statistics (percentages, means, standard deviations), as well as statistical and clinical change. Qualitative in-depth interviews will be analyzed using thematic content analysis.

Plan for activities and dissemination:

Scheduled start of data collection is September 2020. The data collection will continue until the summer of 2021. The follow-up period will be completed by the end of 2021.

The results of the feasibility study will be published in peer-reviewed journals. Furthermore, the results will be disseminated to the public through media (including social media), and as information aimed at both health and social care professionals, patient groups and user forums.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* access to the Internet
* interested in receiving Internet treatment for changing drinking habits
* a score of 6 or higher for women and 8 or higher for men on the Alcohol Use Disorder Identification Test (AUDIT)

Exclusion Criteria:

* diagnosed alcohol dependence or addiction to other drugs and already in treatment
* serious reading and/or writing difficulties
* cognitive impairment/dementia
* severe mental disorder or in need of other treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
The Alcohol Use Disorders Identification Test (AUDIT) | AUDIT will measure whether there is a change in alcohol intake during the treatment period (8-12 weeks) and at follow-up (6 months after the end of treatment).
  AUDIT is a screening instrument consisting of 10 questions designed to identify hazardous (risky) and harmful use of alcohol in adults. Based on the 10 questions, a score is calculated indicating whether the person is at risk for developing more serious alcohol problems. A cut-off score of > 6 points indicates risky use in women, and a cut-off score of > 8 points indicates risky use in men.
The Timeline Followback (TLFB) for alcohol | TLFB will calculate the intake of alcohol units (AE) and change in the seven-day period from the first assessment to the 6 months follow-up.
  TLFB for alcohol is an assessment tool that includes estimates of daily alcohol intake over a specific period, e.g. within seven days. TLFB provides information on various dimensions of the person's drinking habits, such as the number of drinking days and the maximum amount of alcohol consumed.

SECONDARY OUTCOMES:
The Drug-Taking Confidence Questionnaire (DTCQ). | DTCQ will measure changes during the treatment course of 8-12 weeks, and at 6 months follow-up.
  DTCQ measures the person's confidence in his or her abilities to cope in situations that are high-risk for substance use. The tool yields information about client strengths and needs in the area of relapse potential in 50 different risk situations.
Symptom Checklist -10 (SCL-10) | SCL-10 will measure changes in psychological distress during the treatment course of 8-12 weeks, and at 6 months follow-up.
  SCL-10 is a self-report questionnaire for identifying symptoms of psychological distress over the past seven days. SCL-10 contains 10 statements.
Patient Health Questionnaire, PHQ-9 | Patient Health Questionnaire (PHQ-9) will measure changes in symptoms of depression during the treatment course of 8-12 weeks, and at 6 months follow-up.
  Patient Health Questionnaire (PHQ-9) consists of nine items and measures key symptoms of depression.
General Anxiety Disorder (GAD-7). | GAD-7 will measure changes in symptoms of anxiety during the treatment course of 8-12 weeks, and at 6 months follow-up.
  GAD-7 is a screening instrument that consists of seven items and measures key symptoms of anxiety.
EuroQol five-dimensional (EQ-5D) descriptive system (EQ-5D-5L) | EQ-5D-5L will measure changes in health-related quality of life during the treatment course of 8-12 weeks, and at 6 months follow-up.
  EQ-5D-5L measures health-related quality of life in five areas; mobility, personal care, activities of daily living, pain/discomfort and anxiety / depression

OTHER OUTCOMES:
Qualitative interviews | Qualitative interviews will be conducted at the end of treatment, immediately after 8-12 weeks completed treatment
  Qualitative interviews will investigate participants' expectations and experience of the intervention, focusing on both the technical solutions related to the intervention and the importance of therapist support.

CONTACTS AND LOCATIONS:
Overall Officials: Else Marie Løberg, PhD, Study Director — Haukeland University Hospital
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Vestfold Hospital, Tønsberg

IPD SHARING:
Plan to Share IPD: No